CLINICAL TRIAL: NCT04140682
Title: Comparison of Proportional Assisted Ventilation and Pressure Support Ventilation in Adult Patients With Prolonged Mechanical Ventilation: A Randomized Controlled Trial
Brief Title: Proportional Assisted Ventilation and Pressure Support Ventilation in Adult Patients With Prolonged Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Chiu-Fan Chen, Principal Investigator, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS99-CT14-15
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Respiratory Failure; Respiration, Artificial
Keywords: Proportional assist ventilation; Pressure support ventilation; Weaning; Prolonged mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAV+ mode (Experimental): Weaning with PAV+ mode
  Interventions: Device: PAV+ mode
- PSV mode (Active Comparator): Weaning with PSV mode
  Interventions: Device: PSV mode

INTERVENTIONS:
Device: PAV+ mode — PAV+ mode by using Puritan-Bennett 840 ventilator
  Arms: PAV+ mode
Device: PSV mode — PSV mode by using Puritan-Bennett 840 ventilator
  Arms: PSV mode

SUMMARY:
A prospective randomized controlled trial was conducted to collect patients with prolonged mechanical ventilation. Patients were randomly assigned to receive PAV+ or PSV as weaning mode. Weaning outcomes were compared between 2 groups.

DETAILED DESCRIPTION:
Pressure support ventilation (PSV) the most frequently used mode of ventilator support in intensive care units, but has several demerits. Proportional assist ventilation with load-adjustable gain factors (PAV+) is a promising mode with better patient synchrony and weaning advantages. However, weaning outcome of PAV+ in patients with prolonged mechanical ventilation has not been evaluated before. We conducted a prospective randomized controlled trial in a tertiary medical center. This study aimed to compare the effectiveness between PAV+ and PSV for weaning adult patients with prolonged mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prolonged mechanical ventilation and transfer to respiratory care center, age of 20 years or older, at least 1 time of extubation failure or spontaneous breathing trial failure in ICU, stable hemodynamics, no vasopressor use, FiO2 = 0.40 or less, external positive end-expiratory pressure = 5 cmH2O or less, PaO2 > 60 mmHg, and body temperature < 38ºC (within 24 hours).

Exclusion Criteria:

* Patients with bronchopleural fistulas, central neurological disorders, hemodialysis, and those with pressure support level already < 15 cmH2O.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2011-04-30 (Actual); Study Completion 2011-04-30 (Actual)

PRIMARY OUTCOMES:
28-day weaning success rate | 28 days
  Weaning success was defined as being alive and liberation from MV for more than 48 hours.

SECONDARY OUTCOMES:
Weaning duration | up to 28 days
  Weaning duration was defined as the time from randomization to successful liberation from MV. For those who failed to liberate from MV throughout the course of weaning trial, the weaning duration was defined from randomization to the end of study (up to 28 days).
Hospital length of stay | up to 123 days
  Patients were followed to discharge to calculate the length of hospitalization
Weaning success at discharge | up to 123 days
  Patients were followed to discharge to calculate weaning success rate at discharge, which is defined as status of being alive and successful weaned at patient discharge
Hospital mortality | up to 123 days
  Patients were followed to discharge to calculate the mortality rate during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Chiu-Fan Chen, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No